CLINICAL TRIAL: NCT02482480
Title: Effects of a Comprehensive Management Program for the Treatment of Obstructive Sleep Apnea Syndrome
Brief Title: Comprehensive Management for the Treatment of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Jose M. Montserrat, MD, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEPAR-ALAT-2014
Record Dates: First submitted 2015-03-25; First posted 2015-06-26 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: SLEEP APNEA SYNDROME
Keywords: SLEEP; APNEA; EXERCISE
MeSH Terms: conditions — Sleep Apnea Syndromes; Apnea; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional group (Experimental): Participants followed a 8-week intervention program with a total of 24 sessions (12 of those were supervised). The aim of the supervision was to increase the adherence to the treatment and to control the compliance of patients. General physical activity consisted in walking along previously standardized urban parks designed for the urban EPOC training project (Arbillaga-Etxarri et al, 2016). The duration of walking were 30 minutes. The physiotherapist supervised the accomplishment of other activities such as oropharyngeal exercises and diet control.
  Oropharyngeal exercises:
  1. Expiratory muscle strength training (EMST):
  2. Masako Manoeuvre
  3. Shaker Head Lift:
  4. Facial exercise
  Interventions: Other: Exercise
- Control Group (Sham Comparator): Control group participants only received general recommendations regarding general physical activity, diet and sleep hygiene. After 8-weeks of control, they were re-evaluated with the same evaluation test used in the beginning of the study period. Recommendations for general physical activity were walking during 30 minutes at least 3 times a week maintaining the greatest possible pace. Also, control group patients received the same diet control document as intervention group and verbal advice for sleep hygiene. Approximately 1 month after enrolment, a follow-up phone call was completed were we also informed about the new re-evaluation data.
  Interventions: Other: Control

INTERVENTIONS:
Other: Exercise — Walking in community Oropharyngeal exercises Diet recommendations Dietary recommendations Education
  Arms: Interventional group
Other: Control — Dietary and general recommendations
  Arms: Control Group

SUMMARY:
Study objetives : The aim of this study is to assess the impact of a combined therapy treatment (physical exercise, oropharyngeal exercises and dietary recommendations) on symptoms and quality of life in patients with OSAS, as an alternative or addition to therapeutic treatment with nocturnal CPAP.

DETAILED DESCRIPTION:
The obstructive sleep apnea syndrome (OSAS) is characterized by repetitive obstruction of the upper airway during sleep. OSAS is associated with a wide range of health consequences such as daytime sleepiness, cognitive impairment and metabolic and cardiovascular diseases. In Spain the prevalence of this disease is 3 to 6%, constituting a public health problem. The recommended first line treatment for OSAS is continuous positive pressure airway (CPAP).

Physical exercise has been shown to ameliorate the consequences of OSAS such as cardiovascular disease, glucose intolerance and fatigue. Scientific studies have shown that vigorous physical activity is associated with a decrease in the prevalence of OSAS, improved sleep efficiency and the Epworth Sleepiness Scale.

Moreover, recent evidence has shown that oropharyngeal exercises can be useful in the treatment of OSAS decreasing neck circumference, snoring, subjective sleepiness and AHI as well as improving the quality of life and saturation oxygen.

The 60-70% of patients with OSAS is overweight or obese showing that a high body mass index (BMI) is an independent risk factor for the occurrence of OSAS. Many studies have shown that weight loss is associated with significant reduction in AHI.

However, despite the scientific evidence to justify the inclusion of these modalities, there is no study that has analyzed the impact of performing together all these interventions. It is expected that the combination can produce a cumulative effect that impacts significantly on improving indicators of OSAS.

The investigators will include patients with a recent diagnosis of moderate or severe OSA. Patients will be randomized to interventional or control group.

Patients included in the study will be followed for almost three months and they will be examined at baseline and after time of follow-up or intervention.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe Obstructive Sleep Apnea Hypopnea Syndrome (AHI > 15/h)

Exclusion Criteria:

* BMI > 40
* Concomitant heart disease, stroke or severe neuromuscular with medical judgment not doing exercise.
* Musculoskeletal disorders that impede the realization of the exercises
* Sleepiness affects your physical or occupational functioning.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Apnea-hipopnea index (AHI) | 10 weeks

SECONDARY OUTCOMES:
OSA symtoms and quality of life | 10 weeks
  Epworth Sleepiness Score (ESE)-Quebec sleep questionnaire (QSQ)
Minutes per day of moderate-to-vigorous physical activity with Sensewear Armband | 10 weeks
Distance walking in the Six minute walking Test | 10 weeks
Anxiety and depression on the Hospital Anxiety and Depression questionnaire | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Torres, MSc, Principal Investigator — University of Barcelona
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes